CLINICAL TRIAL: NCT07191769
Title: The Effect of the Selected Anaesthesia Method on Morbidity and Mortality in Frail Patients Scheduled for Transurethral Surgery
Brief Title: The Importance of Anesthesia Method in Fragile Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: SBU-ANESTEZİ-DMY-04
Record Dates: First submitted 2025-09-09; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Frail Elderly Syndrome
Keywords: frail patient; general anaesthesia; regional anaesthesia
MeSH Terms: interventions — Anesthesia, General; Anesthesia, Conduction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients undergoing general anaesthesia: Patients aged 65 years and older who are scheduled for transurethral surgery, meet frailty criteria, and have an American Society of Anesthesiologists (ASA) physical status classification of I-III will be included in this group after being enrolled in the study and undergoing general anaesthesia.
  Interventions: Procedure: general anaesthesia
- Patients undergoing regional anaesthesia: Patients aged 65 years and older who are scheduled for transurethral surgery, meet frailty criteria, and have an American Society of Anesthesiologists (ASA) physical status classification of I-III will be included in this group after being enrolled in the study and undergoing regional anaesthesia.
  Interventions: Procedure: regional anaesthesia

INTERVENTIONS:
Procedure: general anaesthesia — Patients undergoing general anaesthesia
  Groups: Patients undergoing general anaesthesia
Procedure: regional anaesthesia — Patients undergoing regional anaesthesia
  Groups: Patients undergoing regional anaesthesia

SUMMARY:
The aim of this study is to comparatively evaluate the effects of different anaesthesia methods (spinal anaesthesia and general anaesthesia) administered to frail elderly patients scheduled for transurethral surgery (e.g. TUR-Prostate or TUR-Bladder) on postoperative morbidity and mortality rates.

DETAILED DESCRIPTION:
When planning transurethral surgery in frail patients, optimising the anaesthesia method is critical in minimising perioperative risks. In a 2021 study by Darwish et al. (1), 28,486 TUR-P cases were grouped according to the selected anaesthesia method. The 30-day mortality rate was 0.4% in the neuroaxial anaesthesia (spinal/epidural) group and 0.7% in the general anaesthesia group; the neuroaxial anaesthesia group showed significantly better outcomes in terms of secondary morbidity rates such as mortality and sepsis. However, there are studies in the literature supporting general anaesthesia. A study by Ayoub et al. (4) emphasised that in frail patients, similar morbidity rates can be achieved with general anaesthesia or spinal anaesthesia; spinal anaesthesia may increase the risk of hypotension and bradycardia. Based on these studies, the selection of the appropriate anaesthesia method for transurethral procedures is of critical importance in terms of patient morbidity and mortality rates. This study aims to contribute to clinical guidelines by clarifying which type of anaesthesia is safer in this specific demographic and clinical group. Within the scope of the research, parameters such as complications associated with the anaesthesia method, length of hospital stay, readmission rate, and 30-day mortality are analysed with the aim of determining the most appropriate and safest anaesthesia method for the vulnerable patient group.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients aged 65 and over
* ASA (American Society of Anaesthesiologists) physical condition classification I-III patients
* meeting the criteria for frailty

Exclusion Criteria:

* Non-elective emergency surgeries
* Patients under 65 years of age
* Patients classified as ASA Class IV
* Patients unable to provide informed consent due to cognitive impairment
* Patients who have previously undergone major neurological or cardiac surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 65 years and older who are scheduled for transurethral surgery (such as TUR-P or TUR-M), meet frailty criteria, and have an American Society of Anesthesiologists (ASA) physical status classification of I-III will be included in the study. A validated frailty score (FRAIL Survey) will be used for frailty assessment.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Postoperative morbidity | 30-day postoperative morbidity
  Morbidity rates up to the 30th day postoperatively will be recorded. Patients will be contacted by phone and the data will be recorded.
Postoperative mortality | 30-day postoperative mortality
  Mortality rates up to the 30th day postoperatively will be recorded. Patients will be contacted by phone and the data will be recorded.

SECONDARY OUTCOMES:
intraoperative complications, | perioperative period
  In the study, complications that develop during surgery (arrhythmia etc.), whether the surgical time differs between the two groups, and the length of hospital stay will be recorded.
Duration of surgery | Until the end of the surgery
  The surgical durations of patients in both groups will be recorded in the study.
Length of hospital stay | first week after surgery
  The length of time the patient stays in hospital for the operation will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Yamac, Principal Investigator — Sultan Abdülhamid Han education and research hospital

IPD SHARING:
Plan to Share IPD: No